CLINICAL TRIAL: NCT06968442
Title: SARS-CoV-2 Antibody-mediated Inflammatory Responses by Macrophages in Individuals With and Without Obesity
Brief Title: The Role of Obesity in Severe COVID-19 Pathophysiology
Acronym: SAMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Franciscus Gasthuis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL88800.100.25
Record Dates: First submitted 2025-04-28; First posted 2025-05-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: COVID-19; Antibody COVID-19
Keywords: COVID-19; Obesity; Antibodies; Macrophages; Immunity; Fc receptors
MeSH Terms: conditions — COVID-19; Obesity | interventions — Phlebotomy; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: The investigators include a cohort of obesity patients (all BMI >35) who are eligible for bariatric surgery and a control cohort of age and sex matched lean (all BMI <25) healthcare workers. From all individuals, blood is collected and immunological analyses are performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- General (Other): The intervention is a blood collection, whereafter blood will be analyzed for immunological parameters.
  Interventions: Procedure: Venipuncture

INTERVENTIONS:
Procedure: Venipuncture — Simple blood collection
  Other Names: Venapuncture; Blood collection

SUMMARY:
The coronavirus disease 2019 (COVID-19) pandemic, caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), has resulted in millions of deaths worldwide. As of 2024, the SARS-CoV-2 Omicron variant is the predominant strain circulating within the population, generally causing mild upper respiratory tract infections. However, hospitalizations and case fatalities due to COVID-19 continue, and there is a high probability that a new human coronavirus will emerge in the future. Understanding the pathophysiology of severe COVID-19 remains highly relevant, as its mechanisms may be comparable to those of other respiratory viral infections.

SARS-CoV-2 infects human cells primarily by binding to angiotensin-converting enzyme 2 (ACE2) and type 2 transmembrane serine protease (TMPRSS2) receptors, which are both expressed in alveolar epithelial type II cells, through the virus' spike protein. In a later stage, the replication of SARS-CoV-2 and activation of resident immune cells lead to the infiltration and activation of large numbers of innate immune cells. Consequently, this results in an excessive pro-inflammatory immune response, including increased production of IL-6, a hallmark cytokine of severe COVID-19. Eventually, the excessive inflammation results in microthrombus formation and pulmonary edema.

Further studies have indicated that SARS-CoV-2 spike-specific antibodies, along with alveolar macrophages, play a pivotal role in the pathophysiology of severe COVID-19. Alveolar macrophages, which reside in the lung alveoli, are typically the first immune cells to sense pulmonary pathogens. However, these cells can also bind IgG antibodies through their Fc-receptor, leading to cellular activation. When stimulated with both a viral stimulus and anti-SARS-CoV-2 IgG antibodies from severe COVID-19 patients (a situation similar to that in the lungs of these patients) alveolar macrophages elicit a significant proinflammatory response. This response aligns with the observed post-seral conversion deterioration in COVID-19 patients.

Obesity is a significant risk factor for developing severe COVID-19, but the underlying mechanism is not well understood. Previous studies report that macrophages in obese patients are skewed towards a pro-inflammatory phenotype due to altered fatty acid contents, particularly increased saturated fatty acids. Using our in vitro obesity model, which incorporates higher saturated fatty acid contents, the investigators already demonstrated that SARS-CoV-2 antibody-mediated inflammation of alveolar macrophages is increased (unpublished data). Thus, this may explain why obese patients are more likely to develop severe COVID-19.

To validate these in vitro findings, the investigators aim to confirm these results in monocyte-derived macrophages isolated from individuals with and without obesity. Additionally, the investigators will investigate the underlying mechanisms involved in detail. This study will provide valuable insights into the role of obesity in severe COVID-19 and potentially inform therapeutic strategies for at-risk populations.

DETAILED DESCRIPTION:
This is a mono-center, prospective cohort study involving both a test group and a control group. The test group comprises patients with obesity eligible for bariatric surgery at Franciscus Hospital, while the control group consists of age- (maximum 5-year difference) and sex-matched non-obese healthcare workers at Franciscus Hospital. Blood samples will be collected from all participants at a single time point.

Obese patients will be approached for informed consent during their intake appointments, typically weeks to months before their bariatric surgery. Blood samples will be collected before surgery or during surgery to minimize any potential adverse effects. Collaborating researchers from the surgery department will manage the inclusion of obese patients and coordinate their blood collection.

For the non-obese control group, investigators from MMI will manage participant inclusion and blood sample collection.

Participants from Franciscus Hospital with obesity (Cohort 1) and healthcare workers without obesity (Cohort 2) will undergo a single venipuncture after an 8-hour fasting period. A total of 40 mL of blood will be collected in four 10 mL EDTA tubes.

At the Medical Microbiology and Infection Control (MMI) laboratory of Franciscus, blood samples will be collected after which these are sent to the Center for Infection and Molecular Medicine (CIMM) laboratory in Amsterdam UMC. Here, blood will be processed (i.e., isolation of plasma, monocytes, and remaining peripheral blood mononuclear cells (PBMCs)), where after monocytes will be put into culture to become monocyte-derived macrophages. Macrophage stimulations and additional macrophage analyses will be performed at Amsterdam UMC. Data obtained from analyses in Amsterdam UMC will be further analyzed in Amsterdam UMC by coordinating investigator Ashwin Mak (who is also affiliated at CIMM in Amsterdam UMC) and co-investigator Dr. Jeroen den Dunnen. Monocytes and plasma will be stored in Amsterdam UMC until the end of this study, where after the remaining materials will be transported to Franciscus.

Isolated PBMCs and plasma will be transported in the following days after isolation to Franciscus MMI for T cell stimulations and antibody analyses. In the analyses overview below, the location where each analysis will be performed is noted (i.e., MMI and CIMM). Coded samples and data will be stored at Amsterdam UMC until the end of this study, where after these samples are destroyed and data are deleted. MTA and DTA documents will be prepared for the transfer of blood and data to Amsterdam UMC.

ELIGIBILITY:
Inclusion criteria:

Cohort 1 (obesity cohort)

* ≥18 and ≤65 years of age
* BMI ≥30 kg/m²
* Patient of Franciscus Hospital

Cohort 2 (control cohort)

* ≥18 and ≤65 years of age
* BMI <25 kg/m²
* Healthcare workers of Franciscus Hospital

Exclusion Criteria (for both cohorts):

* Acute infection or current systemic immunological disorders
* Use of immune-modulatory medication (i.e., corticosteroids and biologicals)
* Hormonal therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
The concentration of pro-inflammatory cytokines (IL-6, IL-1β, and TNF) produced by macrophages upon both SARS-CoV-2 viral and antibody costimulation. | Baseline
  Monocytes will be isolated from blood of participants of both groups, whereafter these are differentiated into macrophages. These macrophages will be stimulated with a virus and SARS-CoV-2 IgG combined stimulation. After the stimulation, the concentration of pro-inflammatory cytokines is measured in the supernatant of the macrophages.

SECONDARY OUTCOMES:
The concentration of pro-inflammatory cytokines (IL-6, IL-1β, and TNF) produced by macrophages upon separate viral stimulation or SARS-CoV-2 antibody stimulation | Baseline
  Monocytes will be isolated from blood of participants of both groups, whereafter these are differentiated into macrophages. These macrophages will be stimulated separately with a virus and SARS-CoV-2 IgG stimulation. After the stimulation, the concentration of pro-inflammatory cytokines is measured in the supernatant of the macrophages.
The plasma concentration of pro-inflammatory cytokines | Baseline
  Pro-inflammatory cytokines will be directly measured in plasma.
Measurement of other cytokines that are produced by macrophages upon viral stimulation, antibody stimulation, or both | Baseline
  Monocytes will be isolated from blood of participants of both groups, whereafter these are differentiated into macrophages. These macrophages will be stimulated with a viral stimulation, SARS-CoV-2 IgG stimulation or both combined. After the stimulations, the concentration of additional cytokines (IL-10, IFNg, IFNa, IFNb) will be measured in the supernatant of the macrophages.
Expression levels of Fc receptors on the surface of macrophages | Baseline
  Macrophages will be analyzed by flow cytometry to determine the expression levels of Fc receptors (including CD16, CD32a, CD32b, CD64).
The level of intracellular lipids in monocytes | Baseline
  Monocytes isolated from blood will be analyzed by flow cytometry to assess the intracellular lipid content
Gene expression levels of proteins related to immune signalling or metabolic pathways | Baseline
  Molecular techniques will be applied to assess the gene expression levels of interesting proteins involved in immune signalling or metabolic pathways.
Chromatin accessibility, measured as the number of 'reads per genomic region' of genes related to Fc-receptor activation in macrophages | Baseline
  ATAC-seq will be applied to determine the chromatine accessibility of genes related to Fc-receptor (i.e., receptors binding the Fc-part of antibodies) activation in macrophages. These include genes encoding for the receptors itself, as well as genes encoding for proteins related with the related intracellular signalling pathways upon Fc-receptor activation. The measured unit will be the number of reads per genomc region.
The level of lactate production by macrophages upon stimulation with anti-SARS-CoV-2 IgG. | Baseline
  Lactate is the final product of the glycolysis metabolic pathway. The level of lactate produced by macrophages, thus resembling glycolysis activity, will be assessed after stimulaten with anti-SARS-CoV-2 IgG. The concentration will be measured in mM.
The concentration of proteins in plasma | Baseline
  Using a proteomics approach, the concentration of over 1000 proteins will be assessed in plasma.
The level of SARS-CoV-2 specific T cell responses and plasma antibodies | Baseline
  To determine the adaptive immunity against SARS-CoV-2, T cell responses and antibodies specific to SARS-CoV-2 proteins Spike, Spike S2, Spike S2, and Nucleocapsid will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: David S.Y. Ong, M.D., Ph.D., Pharm.D., M.Sc., Principal Investigator — Franciscus Hospital
Locations (1):
- Franciscus, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
If requested we will make the IPD available

REFERENCES:
- [Background] Hoepel W, Chen HJ, Geyer CE, Allahverdiyeva S, Manz XD, de Taeye SW, Aman J, Mes L, Steenhuis M, Griffith GR, Bonta PI, Brouwer PJM, Caniels TG, van der Straten K, Golebski K, Jonkers RE, Larsen MD, Linty F, Nouta J, van Roomen CPAA, van Baarle FEHP, van Drunen CM, Wolbink G, Vlaar APJ, de Bree GJ, Sanders RW, Willemsen L, Neele AE, van de Beek D, Rispens T, Wuhrer M, Bogaard HJ, van Gils MJ, Vidarsson G, de Winther M, den Dunnen J. High titers and low fucosylation of early human anti-SARS-CoV-2 IgG promote inflammation by alveolar macrophages. Sci Transl Med. 2021 Jun 2;13(596):eabf8654. doi: 10.1126/scitranslmed.abf8654. Epub 2021 May 11. PMID 33979301